CLINICAL TRIAL: NCT02627157
Title: Measurements of Corneal Biomechanical Properties Using a Dynamic Scheimpflug Analyzer for Young Healthy Adults in South Korea
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0944
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- myopia patients: 20 to 40 years of age and have myopia with a spherical equivalent (SE) between 0.00 and -11.00 diopters (D)
  Interventions: Device: Dynamic Scheimpflug Analyzer

INTERVENTIONS:
Device: Dynamic Scheimpflug Analyzer — Measurements of Corneal Biomechanical Properties Using a Dynamic Scheimpflug Analyzer

SUMMARY:
The human cornea is affected by the magnitude and velocity of both internal and external forces because the cornea has both static and dynamic resistance components. Considering these natures of the human cornea, many investigators have tried to demonstrate corneal biomechanical properties to understand these characteristics of the cornea. Corneal biomechanical properties are known to influence the accuracy of measurements in intraocular pressure (IOP) and are recognized as important factor to explain the susceptibility of development of glaucomatous damage. Until recently, the only instrument which enabled the in vivo measurements of the ocular biomechanical properties was ocular response analyzer (ORA, Reichert Ophthalmic Instruments, Depew, NY, USA).8 The ORA has been used to assess the biomechanical properties of the cornea according to the dynamic bidirectional applanation process. A dynamic Scheimpflug analyzer (corneal visualization Scheimpflug technology [Corvis ST], OCULUS, Wetzlar, Germany) has been introduced recently and has become a useful instrument for evaluating corneal biomechanical properties. The dynamic Scheimpflug analyzer captures the dynamic process of corneal deformation caused by an air puff using an ultra-high-speed Scheimpflug camera at a rate of up to 4,330 images per second. Until now, well-organized analysis on the normative data of the corneal biomechanical profiles measured with the dynamic Scheimpflug analyzer for young healthy adults has not been reported yet. Hence, in the present study, we aim to conduct normative data analysis for the corneal biomechanical properties with the dynamic Scheimpflug analyzer in a cohort of young healthy adults in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included in analyses if they are 20 to 40 years of age
* Participants who have myopia with a spherical equivalent (SE) between 0.00 and -11.00 diopters (D)

Exclusion Criteria:

* Participants will be excluded from analyses if they had previous ocular or intraocular surgery, a visual field defect, suspicious optic disc appearance, IOP ≥ 30 mmHg, or presence of corneal abnormalities such as keratoconus and forme fruste keratoconus, corneal scarring that would preclude accurate measurements.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young myopic patients
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
applanation time (AT) | 1 hour
applanation length (AL) | 1 hour
corneal velocity (CV) | 1 hour
deformation amplitude | 1 hour
peak distance | 1 hour
radius | 1 hour
maximal concave power | 1 hour
central corneal thickness (CCT) | 1 hour
intraocular pressure (IOP) | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet